CLINICAL TRIAL: NCT06887634
Title: Rebozo and Maternal Procedures to Reduce Persistent Occiput Posterior Position of the Fetal Head: a Randomized Clinical Trial - the ReMaP-POPP RCT -
Brief Title: Rebozo and Maternal Procedures to Reduce Persistent Occiput Posterior Position of the Fetal Head
Acronym: ReMaP-POPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: Fondazione IRCCS San Gerardo dei Tintori (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID 5499_18.12.2024_M bis
Record Dates: First submitted 2025-03-06; First posted 2025-03-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-03

CONDITIONS: Persistent Occiput Posterior Position During Labor
Keywords: Occiput posterior position; Persistent Occiput Posterior Position; Rebozo technic; Maternal postures

STUDY DESIGN:
Intervention Model Description: pragmatic, open-label, single-center randomized controlled trial with two parallel groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rebozo and Maternal Procedures (Active Comparator): Combination of forward-leaning inversion (FLI) and side-lying release (SLR) and Rebozo technique in a pre-specified order (see Assigned Interventions).
  Interventions: Other: Rebozo and Maternal Procedures
- Control group (Active Comparator): Standard of care, including upright, semi-recumbent, lateral recumbent, and hands-and-knees position.
  Interventions: Other: Control

INTERVENTIONS:
Other: Rebozo and Maternal Procedures — Combination of FLI and side-lying release SLR and Rebozo technique in a pre-specified order:
  1) FLI for 30 seconds repeated for 3 subconsequent contractions; 2) SLR for 30 seconds repeated for 3 consequent contractions; 3) Rest with free maternal postures for 15 minutes; 4) 15 minutes of Rebozo on maternal pelvis (women on hands and knees); 5) Rest with free maternal postures for 15 minutes; 6) 15 minutes of Rebozo on the side of the fetal spine (supine women).
  Duration of the intervention ranges between 90 and 105 minutes. The intervention will start within thirty minutes after randomization; it can be interrupted at any time if needed. It will be considered performed when the proposed sequence is completed. After completion of the sequence, women will be allowed to move freely and adopt different postures. No FLI or SLR procedures or the Rebozo technique will be further allowed until sonographic assessment of the fetal head is performed at 3 hour and thirty after randomization
  Arms: Rebozo and Maternal Procedures
Other: Control — Standard of care, including upright, semi-recumbent, lateral recumbent, and hands-and-knees position. They will not receive forward-leaning inversion (FLI) and side-lying release (SLR) and Rebozo technique. the control group will continue to adopt maternal postures with no possibility of performing the FLI or SLR procedures or the Rebozo technique until sonographic assessment of fetal head position is completed at 3 hours and thirty after randomization.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to assess whether a combination of forward-leaning inversion and side-lying release procedures and Rebozo technique in a pre-specified sequence during the first stage of labor among women with a posterior fetus would favor anterior rotation. The main questions it aims to answer is:

• What is the probability of persistent occiput posterior position of the fetal head three hours and thirty minutes after randomization, diagnosed by sonography? Researchers will compare the intervention group, which received a sequence of forward-leaning inversion (FLI), side-lying release procedures (SLR), and the Rebozo technique (lasting 90-105 minutes), to the control group, which received standard care (free maternal postures), to assess whether the specific combination of interventions in the experimental group reduces the probability of the fetal head remaining in the occiput posterior position.

Participants in the intervention group will undergo a combination of forward-leaning inversion, side-lying release procedures, and the Rebozo technique, administered in a pre-determined sequence. In contrast, participants in the control group will receive standard care (free maternal postures).

ELIGIBILITY:
Inclusion Criteria:

* woman in labor between 3 and 8 cm of cervical dilation
* woman with a singleton term fetus (≥37 0/7 weeks of gestation) in an Occiput Posterior Persistent Position clinically diagnosed and confirmed by transabdominal sonography

Exclusion Criteria:

* Women with growth restricted fetuses according to the Delphi's consensus
* Fetuses with congenital anomalies or infections or with chromosomal abnormalities
* Intrauterine fetal demise
* Fetal and/or maternal conditions requiring urgent or emergent delivery or impeding the use of FLI and SLR and/or the Rebozo technique (non-reassuring fetal heart rate, abnormal vaginal bleeding, immobilizing epidural analgesia, polyhydramnios, extrapelvic fetal head, body mass index ≥35 Kg/m2, hypertensive disorders of pregnancy with inadequate control of blood pressure, maternal heart disease in class III to V according to the modified World Health Organization, glaucoma or ocular surgery, esophageal reflux disease, hypermobile sacro-ileac joint, and severe symphysis dysfunction)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Probability of occiput posterior position of the fetal head three hours and thirty minutes after randomization | Three hours and thirty minutes after randomization. For women who will give birth before the end of the three hours and a half after randomization, fetal head position at birth will be considered as the fetal head position for this outcome
  This outcome will be measured by suprapubic transabdominal sonography by a trained clinician blinded to the randomization group. The fetal head position will be classified into one of three categories: occiput anterior (right and left), occiput transverse (right and left), and occiput posterior (right and left). If fetal head position cannot be clearly defined, sonography will be repeated by another trained, senior clinician. For women who will give birth before the end of the three hours and a half after randomization, fetal head position at birth will be considered as the fetal head position for this outcome.

SECONDARY OUTCOMES:
Probability of occiput posterior position confirmed by ultrasound examination at full cervical dilation | full cervical dilation (before the beginning of active maternal pushing efforts); for women who will give birth before sonography at full dilation can be performed, information regarding fetal head position at this timing will be considered as "missing".
  This outcome will be measured, before the beginning of active maternal pushing efforts, by suprapubic transabdominal sonography by a trained clinician blinded to the randomization group. The fetal head position will be classified into one of three categories: occiput anterior (right and left), occiput transverse (right and left), and occiput posterior (right and left). If fetal head position cannot be clearly defined, sonography will be repeated by another trained, senior clinician. For women who will give birth before sonography at full dilation can be performed, information regarding fetal head position at this timing will be considered as "missing".
Probability of occiput posterior position at delivery | At birth. In women undergoing operative delivery, the fetal head position diagnosed by sonography right before delivery will be considered as the position at birth
  This outcome will be measured by clinical diagnosis at birth. In women undergoing operative delivery, the fetal head position diagnosed by sonography right before delivery will be considered as the position at birth
Duration of labor | From the diagnosis of active first stage of labor up birth.
  This outcome will be measured calculating the time (minutes) between the diagnosis of active first stage of labor and birth.
Mode of delivery | At birth
  This outcome could be measured calculating the probability of experiencing a spontaneous vaginal birth, a vacuum assisted vaginal birth or a caesarean section
Perineal lacerations | At birth
  This outcome will be measured by calculating within women who had spontaneous vaginal birth or vacuum assisted vaginal birth, the probability of having third degree perineal tear, of having fourth degree of perineal tear, of having episiotomy.
Primary postpartum hemorrhage | At birth
  This outcome will be measured by calculating the probability of blood loss ≥1000 mL
Woman's pain intensity and ability to cope with pain | Within 30 minutes after randomization and at 3 hours and thirty minutes after randomization
  This outcome will be measured using the Pain Intensity Scale, ranging from 0 to 10 (0 equal to 'no pain' and 10 equal to 'worst pain imaginable), and the Pain Coping Scale, ranging from 10 to 0 (10 equal to 'no need to cope - very easy' and 0 'totally unable to cope').
Maternal birth satisfaction level | Assessed at least 24 hours after delivery up hospital discharge
  This outcome will be measured using the italian version of "Birth Satisfaction Scale-Revised" (BSS-R), ranging from 0 to 40 (higher scores is associated to higher maternal satisfaction at birth).
Rate of newborn admission to neonatal intensive care unit | Before hospital discharge, up to 5 days postpartum
  This outcome will be measured calculating the probability of neonatal intensive care unit admission until hospital discharge
Rate of pelvic floor and sexual dysfunction | At 6-9 months postpartum
  This outcome will be measured through:
  Pelvic Floor Disability Index (PFDI-20) for pelvic floor dysfunction assessment. It ranges from 0 to 300 and higher scores indicate greater pelvic floor dysfunction and distress.
Rate of pelvic floor and sexual dysfunction | At 6-9 months postpartum
  This outcome will be measured through:
  Validated Italian-language questionnaires: Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12, short form) for sexual function assessment. It ranges from 0 to 48 and higher scores indicate better sexual function.
Rate of pelvic floor and sexual dysfunction | At 6-9 months postpartum
  This outcome will be measured through:
  - Pelvic Organ Prolapse Quantification (POP-Q) score to evaluate prolapse severity. It ranges from 0 stage to IV stage and higher stages indicate more severe pelvic organ prolapse.
Rate of pelvic floor and sexual dysfunction | At 6-9 months postpartum
  This outcome will be measured through:
  - Modified Oxford Grading System. It ranges from 0 to 5 and higher scores indicate better muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ornaghi, PHD, Principal Investigator — School of Medicine and Surgery, University of Milano-Bicocca, 20900 Monza, Italy
Locations (1):
- IRCCS San Gerardo dei Tintori, Monza, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, the data dictionary, and statistical analysis code will be made available upon reasonable request after publication of the primary results. Materials related to the intervention (including any instructional tools used in the trial) will also be shared if applicable. Data access will require submission of a brief proposal outlining the intended use, which will be reviewed by the study team. Approved data will be shared via secure data transfer platforms. Consent for future data sharing will be obtained from all participants at the time of enrollment. No commercial use of the data will be permitted.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: After the first publication of the primary results up to 5 years
Access Criteria: Data access will be permitted upon submission of a brief proposal outlining the intended use, which will be reviewed by the study team.

REFERENCES:
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Butcher NJ, Monsour A, Mew EJ, Chan AW, Moher D, Mayo-Wilson E, Terwee CB, Chee-A-Tow A, Baba A, Gavin F, Grimshaw JM, Kelly LE, Saeed L, Thabane L, Askie L, Smith M, Farid-Kapadia M, Williamson PR, Szatmari P, Tugwell P, Golub RM, Monga S, Vohra S, Marlin S, Ungar WJ, Offringa M. Guidelines for Reporting Outcomes in Trial Reports: The CONSORT-Outcomes 2022 Extension. JAMA. 2022 Dec 13;328(22):2252-2264. doi: 10.1001/jama.2022.21022. PMID 36511921
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Obstet Gynecol. 2010 May;115(5):1063-1070. doi: 10.1097/AOG.0b013e3181d9d421. No abstract available. PMID 20410783
- [Background] Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 183: Postpartum Hemorrhage. Obstet Gynecol. 2017 Oct;130(4):e168-e186. doi: 10.1097/AOG.0000000000002351. PMID 28937571
- [Background] Menard MK, Main EK, Currigan SM. Executive summary of the reVITALize initiative: standardizing obstetric data definitions. Obstet Gynecol. 2014 Jul;124(1):150-153. doi: 10.1097/AOG.0000000000000322. PMID 24901267
- [Background] Higgins RD, Saade G, Polin RA, Grobman WA, Buhimschi IA, Watterberg K, Silver RM, Raju TNK; Chorioamnionitis Workshop Participants. Evaluation and Management of Women and Newborns With a Maternal Diagnosis of Chorioamnionitis: Summary of a Workshop. Obstet Gynecol. 2016 Mar;127(3):426-436. doi: 10.1097/AOG.0000000000001246. PMID 26855098
- [Background] Frawley H, Shelly B, Morin M, Bernard S, Bo K, Digesu GA, Dickinson T, Goonewardene S, McClurg D, Rahnama'i MS, Schizas A, Slieker-Ten Hove M, Takahashi S, Voelkl Guevara J. An International Continence Society (ICS) report on the terminology for pelvic floor muscle assessment. Neurourol Urodyn. 2021 Jun;40(5):1217-1260. doi: 10.1002/nau.24658. Epub 2021 Apr 12. PMID 33844342
- [Background] Santoro GA, Wieczorek AP, Dietz HP, Mellgren A, Sultan AH, Shobeiri SA, Stankiewicz A, Bartram C. State of the art: an integrated approach to pelvic floor ultrasonography. Ultrasound Obstet Gynecol. 2011 Apr;37(4):381-96. doi: 10.1002/uog.8816. PMID 20814874
- [Background] Dietz HP. Pelvic floor ultrasound: a review. Am J Obstet Gynecol. 2010 Apr;202(4):321-34. doi: 10.1016/j.ajog.2009.08.018. PMID 20350640
- [Background] Dietz HP. Ultrasound imaging of the pelvic floor. Part I: two-dimensional aspects. Ultrasound Obstet Gynecol. 2004 Jan;23(1):80-92. doi: 10.1002/uog.939. PMID 14971006
- [Background] Dietz HP. Pelvic Floor Ultrasound: A Review. Clin Obstet Gynecol. 2017 Mar;60(1):58-81. doi: 10.1097/GRF.0000000000000264. PMID 28005595
- [Background] Volonte' S, Barba M, Cola A, Marino G, Frigerio M. Italian validation of the short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Int Urogynecol J. 2022 Nov;33(11):3171-3175. doi: 10.1007/s00192-022-05235-0. Epub 2022 Jun 1. PMID 35648181
- [Background] Ferreira CH, Barbosa PB, de Oliveira Souza F, Antonio FI, Franco MM, Bo K. Inter-rater reliability study of the modified Oxford Grading Scale and the Peritron manometer. Physiotherapy. 2011 Jun;97(2):132-8. doi: 10.1016/j.physio.2010.06.007. Epub 2010 Oct 22. PMID 21497247
- [Background] Barba M, Cola A, Melocchi T, Braga A, Castronovo F, Manodoro S, Pennacchio M, Munno GM, Ruffolo AF, Degliuomini RS, Salvatore S, Torella M, Frigerio M. Italian validation of the Pelvic Floor Distress Inventory (PFDI-20) questionnaire. Int Urogynecol J. 2023 Oct;34(10):2459-2465. doi: 10.1007/s00192-023-05572-8. Epub 2023 May 17. PMID 37195425
- [Background] Nespoli A, Colciago E, Fumagalli S, Locatelli A, Hollins Martin CJ, Martin CR. Validation and factor structure of the Italian version of the Birth Satisfaction Scale-Revised (BSS-R). J Reprod Infant Psychol. 2021 Nov;39(5):516-531. doi: 10.1080/02646838.2020.1836333. Epub 2020 Oct 21. PMID 33084372
- [Background] Simkin P. Pain, suffering, and trauma in labor and prevention of subsequent posttraumatic stress disorder. J Perinat Educ. 2011 Summer;20(3):166-76. doi: 10.1891/1058-1243.20.3.166. PMID 22654466
- [Background] Barrowclough J, Crowther C, Kool B. Midwives' views on the acceptability of a future trial of the Sims posture for fetal malposition in labor in the context of their knowledge and practice: A mixed-methods study. Eur J Midwifery. 2022 Aug 1;6:50. doi: 10.18332/ejm/150377. eCollection 2022. PMID 35974715
- [Background] Ornaghi S, Bellante N, Abbamondi A, Maini M, Cesana F, Trabucchi M, Corsi D, Arosio V, Mariani S, Scian A, Colciago E, Lettino M, Vergani P. Cardiac and obstetric outcomes in pregnant women with heart disease: appraisal of the 2018 mWHO classification. Open Heart. 2022 Mar;9(1):e001947. doi: 10.1136/openhrt-2021-001947. PMID 35332050
- [Background] Brown MA, Magee LA, Kenny LC, Karumanchi SA, McCarthy FP, Saito S, Hall DR, Warren CE, Adoyi G, Ishaku S; International Society for the Study of Hypertension in Pregnancy (ISSHP). The hypertensive disorders of pregnancy: ISSHP classification, diagnosis & management recommendations for international practice. Pregnancy Hypertens. 2018 Jul;13:291-310. doi: 10.1016/j.preghy.2018.05.004. Epub 2018 May 24. No abstract available. PMID 29803330
- [Background] Rozenberg P, Porcher R, Salomon LJ, Boirot F, Morin C, Ville Y. Comparison of the learning curves of digital examination and transabdominal sonography for the determination of fetal head position during labor. Ultrasound Obstet Gynecol. 2008 Mar;31(3):332-7. doi: 10.1002/uog.5267. PMID 18307213
- [Background] Ghi T, Eggebo T, Lees C, Kalache K, Rozenberg P, Youssef A, Salomon LJ, Tutschek B. ISUOG Practice Guidelines: intrapartum ultrasound. Ultrasound Obstet Gynecol. 2018 Jul;52(1):128-139. doi: 10.1002/uog.19072. PMID 29974596
- [Background] Fulbrook P, Mooney S. Care bundles in critical care: a practical approach to evidence-based practice. Nurs Crit Care. 2003 Nov-Dec;8(6):249-55. doi: 10.1111/j.1362-1017.2003.00039.x. PMID 14725390
- [Background] Crunden E, Boyce C, Woodman H, Bray B. An evaluation of the impact of the ventilator care bundle. Nurs Crit Care. 2005 Sep-Oct;10(5):242-6. doi: 10.1111/j.1362-1017.2005.00134.x. PMID 16161379
- [Background] Donati S, Buoncristiano M, Lega I, D'Aloja P, Maraschini A; ItOSS working group. The Italian Obstetric Surveillance System: Implementation of a bundle of population-based initiatives to reduce haemorrhagic maternal deaths. PLoS One. 2021 Apr 23;16(4):e0250373. doi: 10.1371/journal.pone.0250373. eCollection 2021. PMID 33891629
- [Background] de Wolff MG, Ladekarl M, Sparholt L, Lykke JA. Rebozo and External Cephalic Version in breech presentation (RECEIVE): A randomised controlled study. BJOG. 2022 Sep;129(10):1666-1675. doi: 10.1111/1471-0528.17111. Epub 2022 Mar 8. PMID 35114058
- [Background] Iversen ML, Midtgaard J, Ekelin M, Hegaard HK. Danish women's experiences of the rebozo technique during labour: A qualitative explorative study. Sex Reprod Healthc. 2017 Mar;11:79-85. doi: 10.1016/j.srhc.2016.10.005. Epub 2016 Oct 31. PMID 28159133
- [Background] Cohen SR, Thomas CR. Rebozo Technique for Fetal Malposition in Labor. J Midwifery Womens Health. 2015 Jul-Aug;60(4):445-51. doi: 10.1111/jmwh.12352. PMID 26255805
- [Background] Tully G. Posterior Perspective. Midwifery Today Int Midwife. 2015 Summer;(114):8-11. No abstract available. PMID 26281517
- [Background] Lepleux F, Hue B, Dugue AE, Six T, Riou C, Dreyfus M. [Obstetric data in a population with postural changes during labor and delivery]. J Gynecol Obstet Biol Reprod (Paris). 2014 Sep;43(7):504-13. doi: 10.1016/j.jgyn.2013.06.013. Epub 2013 Aug 22. French. PMID 23972772
- [Background] Lee N, Munro V, Oliver K, Flynn J. Maternal positioning with flexed thighs to correct foetal occipito-posterior position in labour: A systematic review and meta-analysis. Midwifery. 2021 Aug;99:103008. doi: 10.1016/j.midw.2021.103008. Epub 2021 Apr 20. PMID 33895659
- [Background] Liu LP, Chen JH, Yang ZJ, Zhu J. Corrective effects of maternal extreme flexure and hip abduction combined with contralateral side-lying on persistent foetal occipito-posterior position. Int J Nurs Pract. 2018 Oct;24(5):e12663. doi: 10.1111/ijn.12663. Epub 2018 Jun 8. PMID 29882264
- [Background] Bahmaei K, Iravani M, Moosavi P, et al. Effect of maternal positioning with occipito-posterior fetal position during labor on pain intensity and satisfaction of mothers. Iranian Journal of Obstetrics, Gynecology and Infertility 2018;21(5):66-73.
- [Background] Bueno-Lopez V, Fuentelsaz-Gallego C, Casellas-Caro M, Falgueras-Serrano AM, Crespo-Berros S, Silvano-Cocinero AM, Alcaine-Guisado C, Zamoro Fuentes M, Carreras E, Terre-Rull C. Efficiency of the modified Sims maternal position in the rotation of persistent occiput posterior position during labor: A randomized clinical trial. Birth. 2018 Dec;45(4):385-392. doi: 10.1111/birt.12347. Epub 2018 Mar 14. PMID 29537658
- [Background] Ou X, Chen X, Su J. [Correction of occipito-posterior position by maternal posture during the process of labor]. Zhonghua Fu Chan Ke Za Zhi. 1997 Jun;32(6):329-32. Chinese. PMID 9596909
- [Background] Wu X, Fan L, Wang Q. [Correction of occipito-posterior by maternal postures during the process of labor]. Zhonghua Fu Chan Ke Za Zhi. 2001 Aug;36(8):468-9. Chinese. PMID 11758180
- [Background] Molina Reyes C, Munoz-Martinez A, Martiniz-Garcia E, et al. Efficacy of hands and knees maternal posture to correct the occipitoposterior fetal position during labor. index enferm 2014;23:15-20.
- [Background] Guittier MJ, Othenin-Girard V, de Gasquet B, Irion O, Boulvain M. Maternal positioning to correct occiput posterior fetal position during the first stage of labour: a randomised controlled trial. BJOG. 2016 Dec;123(13):2199-2207. doi: 10.1111/1471-0528.13855. Epub 2016 Jan 24. PMID 26806596
- [Background] Stremler R, Hodnett E, Petryshen P, Stevens B, Weston J, Willan AR. Randomized controlled trial of hands-and-knees positioning for occipitoposterior position in labor. Birth. 2005 Dec;32(4):243-51. doi: 10.1111/j.0730-7659.2005.00382.x. PMID 16336365
- [Background] Barth WH Jr. Persistent occiput posterior. Obstet Gynecol. 2015 Mar;125(3):695-709. doi: 10.1097/AOG.0000000000000647. PMID 25730235
- [Background] Andrews CM, Andrews EC. Physical theory as a basis for successful rotation of fetal malpositions and conversion of fetal malpresentations. Biol Res Nurs. 2004 Oct;6(2):126-40. doi: 10.1177/1099800404268318. PMID 15388910
- [Background] Desbriere R, Blanc J, Le Du R, Renner JP, Carcopino X, Loundou A, d'Ercole C. Is maternal posturing during labor efficient in preventing persistent occiput posterior position? A randomized controlled trial. Am J Obstet Gynecol. 2013 Jan;208(1):60.e1-8. doi: 10.1016/j.ajog.2012.10.882. Epub 2012 Oct 26. PMID 23107610
- [Background] Tempest N, Hart A, Walkinshaw S, Hapangama DK. A re-evaluation of the role of rotational forceps: retrospective comparison of maternal and perinatal outcomes following different methods of birth for malposition in the second stage of labour. BJOG. 2013 Sep;120(10):1277-84. doi: 10.1111/1471-0528.12199. Epub 2013 Mar 21. PMID 23906197
- [Background] Stock SJ, Josephs K, Farquharson S, Love C, Cooper SE, Kissack C, Akolekar R, Norman JE, Denison FC. Maternal and neonatal outcomes of successful Kielland's rotational forceps delivery. Obstet Gynecol. 2013 May;121(5):1032-1039. doi: 10.1097/AOG.0b013e31828b72cb. PMID 23635740
- [Background] Le Ray C, Deneux-Tharaux C, Khireddine I, Dreyfus M, Vardon D, Goffinet F. Manual rotation to decrease operative delivery in posterior or transverse positions. Obstet Gynecol. 2013 Sep;122(3):634-40. doi: 10.1097/AOG.0b013e3182a10e43. PMID 23921875
- [Background] Bahl R, Van de Venne M, Macleod M, Strachan B, Murphy DJ. Maternal and neonatal morbidity in relation to the instrument used for mid-cavity rotational operative vaginal delivery: a prospective cohort study. BJOG. 2013 Nov;120(12):1526-32. doi: 10.1111/1471-0528.12398. Epub 2013 Aug 7. PMID 23924292
- [Background] Bertholdt C, Morel O, Zuily S, Ambroise-Grandjean G. Manual rotation of occiput posterior or transverse positions: a systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol. 2022 Jun;226(6):781-793. doi: 10.1016/j.ajog.2021.11.033. Epub 2021 Nov 17. PMID 34800396
- [Background] Blanc J, Castel P, Mauviel F, Baumstarck K, Bretelle F, D'Ercole C, Haumonte JB. Prophylactic manual rotation of occiput posterior and transverse positions to decrease operative delivery: the PROPOP randomized clinical trial. Am J Obstet Gynecol. 2021 Oct;225(4):444.e1-444.e8. doi: 10.1016/j.ajog.2021.05.020. Epub 2021 May 24. PMID 34033811
- [Background] Le Ray C, Serres P, Schmitz T, Cabrol D, Goffinet F. Manual rotation in occiput posterior or transverse positions: risk factors and consequences on the cesarean delivery rate. Obstet Gynecol. 2007 Oct;110(4):873-9. doi: 10.1097/01.AOG.0000281666.04924.be. PMID 17906022
- [Background] Masturzo B, Farina A, Attamante L, Piazzese A, Rolfo A, Gaglioti P, Todros T. Sonographic evaluation of the fetal spine position and success rate of manual rotation of the fetus in occiput posterior position: A randomized controlled trial. J Clin Ultrasound. 2017 Oct;45(8):472-476. doi: 10.1002/jcu.22477. Epub 2017 Apr 3. PMID 28369942
- [Background] Phipps H, Hyett JA, Kuah S, Pardey J, Matthews G, Ludlow J, Narayan R, Santiagu S, Earl R, Wilkinson C, Bisits A, Carseldine W, Tooher J, McGeechan K, de Vries B. Persistent occiput posterior position outcomes following manual rotation: a randomized controlled trial. Am J Obstet Gynecol MFM. 2021 Mar;3(2):100306. doi: 10.1016/j.ajogmf.2021.100306. Epub 2021 Jan 6. PMID 33418103
- [Background] Shaffer BL, Cheng YW, Vargas JE, Caughey AB. Manual rotation to reduce caesarean delivery in persistent occiput posterior or transverse position. J Matern Fetal Neonatal Med. 2011 Jan;24(1):65-72. doi: 10.3109/14767051003710276. Epub 2010 Mar 30. PMID 20350240
- [Background] Elmore C, McBroom K, Ellis J. Digital and Manual Rotation of the Persistent Occiput Posterior Fetus. J Midwifery Womens Health. 2020 May;65(3):387-394. doi: 10.1111/jmwh.13118. Epub 2020 Jun 3. PMID 32491235
- [Background] Le Ray C, Lepleux F, De La Calle A, Guerin J, Sellam N, Dreyfus M, Chantry AA. Lateral asymmetric decubitus position for the rotation of occipito-posterior positions: multicenter randomized controlled trial EVADELA. Am J Obstet Gynecol. 2016 Oct;215(4):511.e1-7. doi: 10.1016/j.ajog.2016.05.033. Epub 2016 May 27. PMID 27242201
- [Background] Levy AT, Weingarten S, Ali A, Quist-Nelson J, Berghella V. Hands-and-knees posturing and fetal occiput anterior position: a systematic review and meta-analysis. Am J Obstet Gynecol MFM. 2021 Jul;3(4):100346. doi: 10.1016/j.ajogmf.2021.100346. Epub 2021 Mar 9. PMID 33705998
- [Background] Hunter S, Hofmeyr GJ, Kulier R. Hands and knees posture in late pregnancy or labour for fetal malposition (lateral or posterior). Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD001063. doi: 10.1002/14651858.CD001063.pub3. PMID 17943750
- [Background] Gardberg M, Tuppurainen M. Anterior placental location predisposes for occiput posterior presentation near term. Acta Obstet Gynecol Scand. 1994 Feb;73(2):151-2. doi: 10.3109/00016349409013418. PMID 8116354
- [Background] Ghi T, Youssef A, Martelli F, Bellussi F, Aiello E, Pilu G, Rizzo N, Frusca T, Arduini D, Rizzo G. Narrow subpubic arch angle is associated with higher risk of persistent occiput posterior position at delivery. Ultrasound Obstet Gynecol. 2016 Oct;48(4):511-515. doi: 10.1002/uog.15808. Epub 2016 Aug 25. PMID 26565728
- [Background] D'Esopo D. The occipito posterior position. Its mechanism and treatment. Am J Obstet Gynecol 1941;42:937-39
- [Background] Longo LD. Classic pages in obstetrics and gynecology. Anatomical variations in the female pelvis and their effect in labor with a suggested classification. William Edgar Caldwell and Howard Carmen Moloy. American Journal of Obstetrics and Gynecology, vol. 26, pp. 479-505, 1933. Am J Obstet Gynecol. 1977 Apr 1;127(7):798. No abstract available. PMID 322490
- [Background] Caughey AB, Sharshiner R, Cheng YW. Fetal malposition: impact and management. Clin Obstet Gynecol. 2015 Jun;58(2):241-5. doi: 10.1097/GRF.0000000000000106. PMID 25851845
- [Background] Le Ray C, Carayol M, Jaquemin S, Mignon A, Cabrol D, Goffinet F. Is epidural analgesia a risk factor for occiput posterior or transverse positions during labour? Eur J Obstet Gynecol Reprod Biol. 2005 Nov 1;123(1):22-6. doi: 10.1016/j.ejogrb.2005.02.009. PMID 16260336
- [Background] Lieberman E, Davidson K, Lee-Parritz A, Shearer E. Changes in fetal position during labor and their association with epidural analgesia. Obstet Gynecol. 2005 May;105(5 Pt 1):974-82. doi: 10.1097/01.AOG.0000158861.43593.49. PMID 15863533
- [Background] Barrowclough JA, Lin L, Kool B, Hofmeyr GJ, Crowther CA. Maternal postures for fetal malposition in labour for improving the health of mothers and their infants. Cochrane Database Syst Rev. 2022 Aug 31;8(8):CD014615. doi: 10.1002/14651858.CD014615. PMID 36043437
- [Background] Badawi N, Kurinczuk JJ, Keogh JM, Alessandri LM, O'Sullivan F, Burton PR, Pemberton PJ, Stanley FJ. Intrapartum risk factors for newborn encephalopathy: the Western Australian case-control study. BMJ. 1998 Dec 5;317(7172):1554-8. doi: 10.1136/bmj.317.7172.1554. PMID 9836653
- [Background] Cheng YW, Shaffer BL, Caughey AB. Associated factors and outcomes of persistent occiput posterior position: A retrospective cohort study from 1976 to 2001. J Matern Fetal Neonatal Med. 2006 Sep;19(9):563-8. doi: 10.1080/14767050600682487. PMID 16966125
- [Background] Pergialiotis V, Bellos I, Fanaki M, Vrachnis N, Doumouchtsis SK. Risk factors for severe perineal trauma during childbirth: An updated meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2020 Apr;247:94-100. doi: 10.1016/j.ejogrb.2020.02.025. Epub 2020 Feb 14. PMID 32087423
- [Background] Foggin HH, Albert AY, Minielly NC, Lisonkova S, Koenig NA, Jacobs EN, Cundiff GW. Labor and delivery outcomes by delivery method in term deliveries in occiput posterior position: a population-based retrospective cohort study. AJOG Glob Rep. 2022 Aug 5;2(4):100080. doi: 10.1016/j.xagr.2022.100080. eCollection 2022 Nov. PMID 36536849
- [Background] Cheng YW, Hubbard A, Caughey AB, Tager IB. The association between persistent fetal occiput posterior position and perinatal outcomes: an example of propensity score and covariate distance matching. Am J Epidemiol. 2010 Mar 15;171(6):656-63. doi: 10.1093/aje/kwp437. Epub 2010 Feb 5. PMID 20139128
- [Background] Cheng YW, Shaffer BL, Caughey AB. The association between persistent occiput posterior position and neonatal outcomes. Obstet Gynecol. 2006 Apr;107(4):837-44. doi: 10.1097/01.AOG.0000206217.07883.a2. PMID 16582120
- [Background] Senecal J, Xiong X, Fraser WD; Pushing Early Or Pushing Late with Epidural study group. Effect of fetal position on second-stage duration and labor outcome. Obstet Gynecol. 2005 Apr;105(4):763-72. doi: 10.1097/01.AOG.0000154889.47063.84. PMID 15802403
- [Background] Ponkey SE, Cohen AP, Heffner LJ, Lieberman E. Persistent fetal occiput posterior position: obstetric outcomes. Obstet Gynecol. 2003 May;101(5 Pt 1):915-20. doi: 10.1016/s0029-7844(03)00068-1. PMID 12738150
- [Background] Fitzpatrick M, McQuillan K, O'Herlihy C. Influence of persistent occiput posterior position on delivery outcome. Obstet Gynecol. 2001 Dec;98(6):1027-31. doi: 10.1016/s0029-7844(01)01600-3. PMID 11755548
- [Background] Parsy T, Bettiol C, Vidal F, Allouche M, Loussert-Chambre L, Guerby P. Persistent occiput posterior position: predictive factors of spontaneous rotation of the fetal head. J Matern Fetal Neonatal Med. 2023 Dec;36(1):2192854. doi: 10.1080/14767058.2023.2192854. PMID 37031965
- [Background] Vitner D, Paltieli Y, Haberman S, Gonen R, Ville Y, Nizard J. Prospective multicenter study of ultrasound-based measurements of fetal head station and position throughout labor. Ultrasound Obstet Gynecol. 2015 Nov;46(5):611-5. doi: 10.1002/uog.14821. PMID 25678449
- [Background] Hjartardottir H, Lund SH, Benediktsdottir S, Geirsson RT, Eggebo TM. When does fetal head rotation occur in spontaneous labor at term: results of an ultrasound-based longitudinal study in nulliparous women. Am J Obstet Gynecol. 2021 May;224(5):514.e1-514.e9. doi: 10.1016/j.ajog.2020.10.054. Epub 2020 Nov 15. PMID 33207231
- [Background] Akmal S, Tsoi E, Howard R, Osei E, Nicolaides KH. Investigation of occiput posterior delivery by intrapartum sonography. Ultrasound Obstet Gynecol. 2004 Sep;24(4):425-8. doi: 10.1002/uog.1064. PMID 15343598
- [Background] Sherer DM, Miodovnik M, Bradley KS, Langer O. Intrapartum fetal head position I: comparison between transvaginal digital examination and transabdominal ultrasound assessment during the active stage of labor. Ultrasound Obstet Gynecol. 2002 Mar;19(3):258-63. doi: 10.1046/j.1469-0705.2002.00641.x. PMID 11896947
- [Background] Sherer DM, Miodovnik M, Bradley KS, Langer O. Intrapartum fetal head position II: comparison between transvaginal digital examination and transabdominal ultrasound assessment during the second stage of labor. Ultrasound Obstet Gynecol. 2002 Mar;19(3):264-8. doi: 10.1046/j.1469-0705.2002.00656.x. PMID 11896948
- [Background] Gardberg M, Tuppurainen M. Persistent occiput posterior presentation--a clinical problem. Acta Obstet Gynecol Scand. 1994 Jan;73(1):45-7. doi: 10.3109/00016349409013392. PMID 8304024
- [Background] Gardberg M, Laakkonen E, Salevaara M. Intrapartum sonography and persistent occiput posterior position: a study of 408 deliveries. Obstet Gynecol. 1998 May;91(5 Pt 1):746-9. doi: 10.1016/s0029-7844(98)00074-x. PMID 9572223
- [Derived] Ornaghi S, Fumagalli S, Antolini L, Panzeri M, Spandrio R, Ferrini S, Nespoli A, Maini M, Locatelli A. Rebozo and maternal postures to prevent persistent occiput posterior position of the fetal head: protocol for a randomised clinical trial 'the ReMaP-POPP RCT'. BMJ Open. 2025 Oct 9;15(10):e103520. doi: 10.1136/bmjopen-2025-103520. PMID 41067764
- See also: National Institute of Health. Racial and Ethnic Categories and Definitions for NIH Diversity Programs and for Other Reporting Purposes 2015 — https://grants-nih-gov.unimib.idm.oclc.org/grants/guide/notice-files/NOT-OD-15-089.html
- See also: ClinicalTrials.gov — https://clinicaltrials.gov/search?cond=fetal%20occiput%20posterior